CLINICAL TRIAL: NCT02831205
Title: Everolimus-Eluting Bioresorbable Scaffolds Versus Everolimus-Eluting Metallic Stents for Diffuse Long Coronary Artery Disease
Acronym: ABSORB-LONG
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to current BVS safety issue
Sponsor: Duk-Woo Park, MD (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Duk-Woo Park, MD, professor of medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2016-14
Record Dates: First submitted 2016-07-06; First posted 2016-07-13 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Percutaneous Transluminal Coronary Angioplasty
Keywords: bioresorbable vascular scaffold; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABSORB BVS (Experimental)
  Interventions: Device: everolimus-eluting bioresorbable vascular (Absorb) scaffold
- XIENCE EES (Active Comparator)
  Interventions: Device: everolimus-eluting cobalt-chromium (Xience) stent

INTERVENTIONS:
Device: everolimus-eluting bioresorbable vascular (Absorb) scaffold
  Other Names: ABSORB BVS
  Arms: ABSORB BVS
Device: everolimus-eluting cobalt-chromium (Xience) stent
  Other Names: XIENCE EES
  Arms: XIENCE EES

SUMMARY:
The purpose of this study is to determine whether ABSORB bioresorbable vascular scaffold is non-inferior to XIENCE everolimus-eluting cobalt-chromium stent with respect to target-lesion failure (TLF) at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and more
* Diffuse long native coronary artery stenosis (>50% by visual estimate) with lesion length of more than 40 mm requiring at least 2 overlapped stents with a reference-vessel diameter of 2.5 to 3.75 mm on visual assessment
* Patients with silent ischemia, stable or unstable angina pectoris, and acute myocardial infarction including NSTEMI or STEMI
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site

Exclusion Criteria:

* Subject has known hypersensitivity or contraindication to device material and its ingredients (everolimus, poly(L-lactide), poly(DL-lactide), lactide, lactic acid) and cobalt, chromium, nickel, platinum, tungsten, acrylic, and fluoro polymers that cannot be adequately premedicated
* Subject has known allergic reaction, hypersensitivity, or contraindication to aspirin; to clopidogrel and prasugrel and ticagrelor; or to heparin and therefore cannot be adequately treated with study medication
* An elective surgical procedure is planned that would necessitate interruption of antiplatelet drugs within 12 m after the procedure
* STEMI requiring primary percutaneous coronary intervention
* Cardiogenic shock
* Restenotic lesions
* Left main
* Extreme angulation (≥90°) or excessive tortuosity (≥two 45° angles) proximal to or within the target lesion
* Heavy calcification proximal to or within the target lesion
* Compromised left ventricular dysfunction (LVEF <30%)
* At the time of screening, the subject has a malignancy that is not in remission
* Terminal illness with life expectancy <1 year
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period
* Patient's pregnant or breast-feeding or child-bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Target lesion failure | 1 year
  event rate for composite of cardiac death, target-vessel myocardial infarction [MI], or ischemia-driven target-lesion revascularization

SECONDARY OUTCOMES:
Cardiac death | 5 years
Target-vessel myocardial infarction | 5 years
Ischemia-driven target-lesion revascularization | 5 years
All-cause mortality | 5 years
event rate of any myocardial infarction; Q-wave vs Non-Q wave, periprocedural myocardial infarction vs follow-up myocardial infarction | 5 years
Any revascularization | 5 years
  Any revascularization; target lesion vs. nontarget lesion, target vessel vs. nontarget vessel, ischemia-driven vs. not ischemia-driven
Target-vessel failure | 5 years
  death from any cause, myocardial infarction, and ischemic-driven target-vessel revascularization
Stent thrombosis | 5 years
event rate of device success or procedural success | 5 years
  Device success defined as angiographic evidence of <30% final residual stenosis of the target lesion.
  Procedural success is defined as mean lesion diameter stenosis ≤50% and without the occurrence of in-hospital myocardial infarction (MI), target vessel revascularization (TVR), or death.
Patient-reported angina status measured by Seattle angina questionnaire | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
This is not a publicly funded trial.